CLINICAL TRIAL: NCT05886205
Title: Exploratory Clinical Study on Induced Pluripotent Stem Cell Derived Exosomes (GD-iEXo-002) Nasal Drops for the Treatment of Refractory Focal Epilepsy
Brief Title: Induced Pluripotent Stem Cell Derived Exosomes Nasal Drops for the Treatment of Refractory Focal Epilepsy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Guidon Pharmaceutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2153-K22C1488
Record Dates: First submitted 2023-05-08; First posted 2023-06-02 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Refractory Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPSC-exosome treatment (Experimental): group1-low-dose group, 8 papatients are treated with 2 μg iPSC-Exos in 200 μL. group2-mid-dose group, 8 papatients are treated with 6 μg iPSC-Exos in 200 μL. group3-mid-dose group, 8 papatients are treated with 18 μg iPSC-Exos in 200 μL. group4-Dose expansion, 10 papatients are treated with iPSC-Exos in 200 μL. iPSC-Exos were administrated for nasal drip, bid for 12 weeks.
  Interventions: Drug: iPSC-Exos

INTERVENTIONS:
Drug: iPSC-Exos — iPSC-Exos were administrated for nasal drip, bid for 12 weeks.

SUMMARY:
Evaluate the safety, tolerability, and preliminary efficacy of GD-iEXo-002 nasal drops in the treatment of focal refractory epilepsy

DETAILED DESCRIPTION:
Epilepsy patients can achieve good control after treatment, but still 30% of patients are medically refractory epilepsy, with the vast majority being focal epilepsy. Recurrent seizures seriously affect the normal development, learning, and life of patients. There is an urgent need for effective drugs to treat refractory focal epilepsy in clinical practice.

Exosomes are a kind of vesicle structures secreted by cells, with a diameter of 30-150 nm, carrying proteins, nucleic acids and other substances. Exosomes have many advantages. As naturally occurring nanoscale secretory membrane vesicles, they have extremely low immunogenicity and good safety, and can cross biological barriers such as the blood-brain barrier and the blood-tumor barrier. Exosomes have specific bioactive substances related to source cells, while stem cell exosomes contain TGF- β、 Functional factors such as BDNF can inhibit cell apoptosis, inhibit inflammatory response, promote angiogenesis, inhibit fibrosis, and enhance tissue repair potential, with a wide range of potential applications.

Induced pluripotent stem cell (iPSC) originates from single cell amplification, with infinite proliferation ability, good consistency and stability; MSCs exhibit significant heterogeneity.

The purpose of this single center, open label clinical trial is to evaluate the safety, tolerability, and preliminary efficacy of induced pluripotent stem cell derived exosomes (iPSC-Exos) nasal drops in the treatment of focal refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. Before conducting this study, understand and sign the informed consent form and comply with the requirements of this study;
2. The subjects are patients with focal epilepsy aged 18 to 70 years (inclusive), regardless of gender;
3. The subjects must comply with the definition of drug resistant epilepsy (ILAE);
4. Subjects must take 1-6 types of anti-epileptic drugs (AEDs), and before entering the screening period, they must take unadjusted types and stable doses of AEDs for at least 4 weeks;
5. Throughout the entire research process, the subject/legal guardian must be able to accurately record the log of epileptic seizures;
6. Subjects must experience at least 4 countable seizures within 28 days prior to the screening period;
7. The subjects are willing and able to comply with the research requirements.

Exclusion Criteria:

1. Unwilling or unable to follow the procedures stipulated in the agreement;
2. Pregnant or lactating women, or women with reproductive potential who are unable or unwilling to take appropriate contraceptive measures;
3. Other uncontrollable diseases that may interfere with the research results, including but not limited to infection, hypertension, diabetes, cardiovascular and cerebrovascular diseases, etc;
4. There are situations that may increase the risk of participating in experiments or research product use, such as liver enzyme elevation exceeding twice the normal upper limit and/or GFR<60 mL/min/1.73 m2;
5. Have a history of drug abuse, alcohol dependence, or smoking within one month;
6. Patients with status epilepticus within one month;
7. Have potential progressive nervous system disease, such as encephalitis, brain tumor, multiple sclerosis or dementia;
8. Patients who plan to undergo epilepsy surgery within six months;
9. Patients with abnormal or diseased nasal structures;
10. Patients with cerebrospinal fluid rhinorrhea;
11. Patients whose family members have not been able to proficiently and correctly master the nasal drip method through standardized training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-05 (Estimated); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
adverse events as assessed by CTCAE | 24 weeks from post-administration
  all potentially treated subjects to assess the safety

SECONDARY OUTCOMES:
Number of participants with abnormal vital signs and abnormal Physical examination findings | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
Number of participants with abnormal Neurological examination | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
  Evaluate general neurological status, muscle strength and tension, sensory ataxia, and pathological signs
Number of participants with abnormal laboratory tests results | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
  Blood routine test, blood biochemistry test ,and electrolytes test
Number of participants with abnormal Urine analysis | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
  Urine routine examination
Seizures frequency | before administration; administration; after the first administration 1 week,2 weeks,4 weeks,8 weeks,12 weeks,16 weeks,24 weeks
  Seizure frequency:
  i. no seizures: any type of seizure disappeared after 28 days of observation; ii. significantly effective: 75%-99% reduction in seizure frequency compared with baseline; iii. Effective: 50%-75% reduction in seizure frequency compared with baseline; iv. Improvement: 25%-50% reduction in the number of seizures compared with baseline, or prolongation, reduction in degree, and shortening of duration between episodes; v. Ineffectiveness and exacerbation: Ineffectiveness refers to a decrease or increase of <25% in the number of seizures compared with baseline, and exacerbation refers to an increase in the frequency of seizures from baseline ≥25%.
Scalp electroencephalogram monitoring | Screening, after the first administration 12 weeks
Head magnetic resonance imaging (MRI) examination | Screening, after the first administration 12 weeks

OTHER OUTCOMES:
Exploratory research-1 | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
  The protein concentration of GFAP, IL-1 β、 IL-6、IL-10、IL-17a、TGF- β、 MCP-1 and TNF- α in blood
Exploratory research-2 | Screening, after the first administration 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 24 weeks
  T cell, B cell, NK cell subpopulation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Han, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li A, Zhao Z, Mi R, Xue G. The Evolving Role of Mesenchymal Stem Cells and Their Exosomes in Epilepsy Management: From Bench to Bedside. Stem Cells Int. 2026 Jan 28;2026:4989846. doi: 10.1155/sci/4989846. eCollection 2026. PMID 41613983